CLINICAL TRIAL: NCT03274154
Title: Efficacy and Tolerance Evaluation of an Anti-age Food Supplement: a Randomized, Controlled Clinical Study Versus Untreated Group
Brief Title: Efficacy and Tolerance Evaluation of an Anti-age Food Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DERMING E0116
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Moderate-severe Skin Aging/Photoaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Hyaluron 465 Innēov (Experimental): 43 caucasian female subjects have taken during a meal, for the first 4 months of trial,1 capsule and 1 tablet/die of the food supplement composed with a precursor of HA (glucosamine) and an enzymatic co-factor of HA synthesis (manganese) .
  Interventions: Dietary Supplement: Pre-Hyaluron 465 Innēov
- Untreated group (No Intervention): 23 caucasian female subjects untreated

INTERVENTIONS:
Dietary Supplement: Pre-Hyaluron 465 Innēov — Food supplement consisting og a tablet and a capsule, composed with a precursor of HA (glucosamine) and an enzymatic co-factor of HA synthesis (manganese)
  Arms: Pre-Hyaluron 465 Innēov

SUMMARY:
Efficacy and Tolerance Evaluation of an Anti-age Food Supplement: a Randomized, Controlled Clinical Study Versus Untreated Group

DETAILED DESCRIPTION:
Aim of the study was to evaluate the anti-age activity of "Pre-Hyaluron 465 Innēov" a food supplement, composed with a precursor of HA (glucosamine) and an enzymatic co-factor of HA synthesis (manganese), taken for 4 consecutive months by female subjects aged 35-60 years (with preference for subjects over 45 years), with moderate-severe skin aging/photoaging according to a reference photographic scale.

The study foresaw the evaluation of the study product activity versus a control group, untreated.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* age 35-60 years (with preference for subjects over 45 years),
* body mass index (BMI) 18-27,
* caucasian healthy subjects with moderate-severe cutaneous aging/photoaging (score > 3 of the reference photographic scale in appendix 8),
* agreeing to present at each study visit without make-up,
* accepting to follow the instructions received by the investigator,
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products,
* agreeing not to apply any topical or take any oral product or nutritional supplementation (vitamins and minerals) other than the investigational products, or use face massages or other means known to improve skin wrinkles or skin qualities during the entire duration of the study,
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study,
* no participation in a similar study actually or during the previous 3 months
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Pregnancy,
* lactation,
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study,
* subjects not in menopause who do not accept to perform the pregnancy test at T0, T1, T2 and T3,
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable.

4.4.2. Dependent on a clinical condition 4.4.2.1. Dermatological disease,

* Presence of cutaneous disease on the tested area as lesions, scars, malformations,
* recurrent facial/labial herpes,
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* Endocrine disease,
* hepatic disorder,
* renal disorder,
* cardiac disorder,
* pulmonary disease,
* cancer,
* neurological or psychological disease,
* inflammatory/immunosuppressive disease,
* drug allergy.
* Anti-inflammatory drugs, anti-histaminic, topic (application on the face) and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of hormonal treatment starting more than 1 year ago),
* assumption of drugs or dietary supplements able to influence the test results in the investigator opinion.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Crow's feet visual score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Wrinkles grade was determined according to l'Oreal clinical standardized photographic scales
Nasolabial folds visual score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Wrinkles grade was determined according to l'Oreal clinical standardized photographic scales
Surface microrelief regularity evaluation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Regularity grade was evaluated according to this score:
  1. = very regular
  2. = regular
  3. = irregular
  4. = very irregular
Skin resistance to pinching clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  The evaluation was performed at level of cheek (malar region) according to the following score: 0 = very important
  1. = important
  2. = moderate
  3. = weak
  4. = very weak
Skin resistance to traction clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  The evaluation was performed at level of cheek (malar region) according to the following score: 0 = very important
  1. = important
  2. = moderate
  3. = weak
  4. = very weak
Skin recovery after pinching clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  The evaluation was performed at level of cheek (malar region) according to the following score: 0 = very important
  1. = important
  2. = moderate
  3. = weak
  4. = very weak
Skin dryness clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Clinical evaluation of skin dryness was performed according to the following score:
  0 = very hydrated skin
  1. = hydrated skin
  2. = normal skin
  3. = kindly dry skin
  4. = dry skin
  5. = very dry skin
Vascular homogeneity clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Homogeneity grade was determined according to specific reference clinical and photographic scales and to the following clinical score:
  0 = very homogeneous
  1. = homogeneous
  2. = quite not homogeneous
  3. = not homogeneous
  4. = very not homogeneous
  5. = marked not homogeneous
Pigmentary homogeneity clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Homogeneity grade was determined according to specific reference clinical and photographic scales and to the following clinical score:
  0 = very homogeneous
  1. = homogeneous
  2. = quite not homogeneous
  3. = not homogeneous
  4. = very not homogeneous
  5. = marked not homogeneous
Skin radiance clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Skin radiance was evaluated using a 10 points scale from very poor to good
Skin plumpness clinical score variation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Skin plumpness was evaluated using a 10 points scale from very poor to good

SECONDARY OUTCOMES:
Superficial skin hydration | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Skin electrical capacitance value measured with Corneometer CM825 (Courage - Khazaka, Köln, Germany).
  The measure of the skin capacitance properties is an indirect expression of its hydration level.
Deep skin hydration | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Tissue dielectric constant value of superficial and deep skin layers measured with MoistureMeterD (Delfin Technologies, Kuopio - Finland)
Determination of roughness profilometric parameters | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  Nasolabial folds profilometric parameters measured by Primos compact portable device (GFMesstechnik). Ra is average roughness of the analysed profile, Rt is wrinkles total high, Rv is wrinkles maximum depth.
Tolerance evaluation | Basal visit (T0), 1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4), 5 months (T5)
  The food supplement tolerance will be evaluated considering: any adverse event related to the study treatment, which occurred during the study; any judgement reported by the volunteers.